CLINICAL TRIAL: NCT05106777
Title: A Multi-center, Open Label Study of Surufatinib in Patients With Osteosarcoma and Soft Tissue Sarcoma
Brief Title: Surufatinib in Patients With Osteosarcoma and Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xing Zhang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-OS101
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib (Experimental): Drug: Surufatinib Surufatinib will be given orally.
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib 300 mg once a day (QD) will be orally administrated on a 21-day cycle.
  Other Names: HMPL-012

SUMMARY:
The purpose is to evaluate the effectiveness and safety of Surufatinib in patients with osteosarcoma and soft tissue sarcoma after Standard chemotherapy therapy.

DETAILED DESCRIPTION:
The study population is patients with advanced osteosarcoma and soft tissue sarcoma who have failed in standard chemotherapy treatment. Surufatinib 300 mg once a day (QD) will be orally administrated on a 21-day cycle. Investigators will evaluate the clinical tumor response to Surufatinib, and if investigators determine that the patient can benefit from the continuation of treatment, the patient will continue the Surufatinib treatment. The duration of study will be 2 years. At the time of study completion, if investigators believe patients can continue to benefit from the investigational product, patients may be provided with Surufatinib with the agreement of the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and voluntarily sign the informed consent form;
2. Male or female, age14-70 years，the body surface area of patients under 18 years old is ≥1.5m2;
3. Histologically or cytologically confirmed advanced osteosarcoma and soft tissue sarcoma (unresectable or metastatic)；
4. The patient had previously failed standard chemotherapy,Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) if 6 months or more have passed since completion of therapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1 (amputation patients 0-2).
6. Life expectancy > 12 weeks.
7. Have measurable disease based on RECIST 1.1.

Exclusion Criteria:

1. Prior treatment with Surufatinib;
2. Systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, and immunotherapy, is planned for the first 4 weeks prior to enrollment or during the study. Radiation radiotherapy (EF-RT) was performed within 4 weeks prior to enrollment.
3. Symptoms that affect oral medication and can not be controlled through proper treatment. (such as inability to swallow, chronic diarrhoea and intestinal obstruction, etc.)
4. With pleural effusion or ascites, cause respiratory syndrome. (> CTC AE grade 2 dyspnea [grade 2 dyspnea refers to shortness of breath during a small amount of activity; affecting instrumental activities of daily life])
5. had central nervous system metastasis;
6. With severe and failed to controlled diseases. (including:1)Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal drug treatment).2)Arrhythmias with grade II and above myocardial ischemia or myocardial infarction, poor control (including corrected QT interval(QTc) men ≥ 450 ms, women ≥ 470 ms) and ≥ 2 congestive heart failure (New York Heart Association ( NYHA) rating).3)Poor control of diabetes (fasting blood glucose > 10mmol / L).4)Active or uncontrolled serious infection (≥ Common Terminology Criteria for Adverse Event(CTC AE) grade 2 infection);5)Patients with active hepatitis B or hepatitis C (hepatitis B: HBsAg-positive and hepatitis B virus(HBV) DNA ≥ 500 IU/mL; hepatitis C: hepatitis C virus(HCV) RNA-positive and abnormal liver function), or active infection requiring antimicrobial treatment (eg Treated with antibacterial drugs, antiviral drugs, antifungal drugs);6)renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;7)Patients with seizures and need treatment.)
7. Accepted surgical treatment, incision biopsy or significant traumatic injury within 28 days before grouping.
8. Participated in other anti-tumor clinical trials within 4 weeks.
9. had other kinds of malignant tumors at the same time; had cardiac insufficiency or arrhythmia;
10. were pregnant or breastfeeding.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free rate at 12weeks | at 12weeks

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
Objective response rate (ORR) | up to 12 months
Disease control rate (DCR) | up to 12 months
Overall survival (OS) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Univerisity, Guangzhou, Guangdong, China